CLINICAL TRIAL: NCT06143189
Title: Well-being Biomarkers and Psychological Functioning of Adult Patients During Chemotherapy Treatment: the Effects of Hospital Clowns and Hosting Conditions
Brief Title: Well-being Biomarkers (BIOSMILE) & Psychology Analyses in Women With Cancer After Hospital Clowns and Hosting Effects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Coimbra (Other)
Collaborators: Portuguese Oncology Institute, Coimbra (Other)
Responsible Party: Principal Investigator, Manuela Grazina, Professor, University of Coimbra
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: BIOSMILE hospital study
Record Dates: First submitted 2023-11-10; First posted 2023-11-22 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Well-Being, Psychological; Biomarkers; Cancer; Ambulatory Care; Complementary Therapies
Keywords: Well-being; biomarkers; BIOSMILE; psychological functioning; ambulatory cancer chemotherapy; hospital clowns
MeSH Terms: conditions — Psychological Well-Being; Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (CG) (Other): Control Group participants were exposed to the normal hosting conditions of the hospital when receiving the usual chemotherapy treatment in ambulatory hospital setting.
  Interventions: Other: Hosting conditions
- Experimental Group (EG) (Experimental): Experimental Group participants were exposed to the Hospital Clowns intervention plus the normal hosting conditions of the hospital when receiving the usual chemotherapy treatment in ambulatory hospital setting.
  Interventions: Other: Hosting conditions; Other: Hospital Clowns

INTERVENTIONS:
Other: Hosting conditions — Hosting conditions care
  the patients are welcome by the nurse, whom talk and give the comfort needed by the patients before starting the treatments.
Other: Hospital Clowns — The HCs "Palhaços D'Opital (PdO)" have a program aiming to bring joy, affection and good mood to adults and elders in hospital environment. They work in pairs, dressed in colorful costumes and they prepared sketches in advance. Their performances recreate day-to-day situations (e.g., clowns trying to install a new TV screen; planning a wedding between the clowns and asking the public for their ideas), ending with specific closure, in order to indicate to the audience that the session had finished and to promote a positive environment after their departure. Each intervention lasted around 15 minutes.
  Arms: Experimental Group (EG)

SUMMARY:
The goal of this interventional study is to evaluate the impact of Hospital Clowns (HCs) intervention, besides to hospital hosting conditions, in the well-being of adult female patients during ambulatory chemotherapy.

The main question[s] it aims to answer are:

* Do the short-term HCs interventions during ambulatory chemotherapy may increase well-being of adult cancer patients in comparison to the hospital hosting conditions?
* Do the short-term HCs interventions, besides the hospital hosting conditions, have effects on well-being biomarkers in association with psychological outcomes?

Participants self-collect a sample of saliva followed by psychological assessment, at a first time-point (basal) and at a final time-point (~after 90 minutes of basal) (pre- and post-test), during the chemotherapy treatment session.

Researchers have compared an HCs intervention plus hosting conditions - experimental group, EG, and hosting conditions only - control group, CG, by the repeated measures of pre- and post-test of biomarkers in saliva and the psychological functioning evaluations, to see the degree of the impact of HCs intervention in the well-being of the patients in comparison with normal hosting conditions. Each HCs intervention lasts around 15 minutes, and it is performed in the middle of the procedure between pre- and post-test.

DETAILED DESCRIPTION:
The recruitment of participants was carried out by a nursing professional in the Portuguese Institute of Oncology of Coimbra, according to the appointments of patients whom would be receiving the usual chemotherapy treatment in ambulatory hospital setting, on the days defined for data and samples collection. Participants were told that they would participate in a study to better understand the variations in the relationships between saliva biomarkers' properties and psychological emotional and attentional states across morning time and those who agree to participate were provided with written informed consent at arrival to ambulatory hospital.

Data were obtained after participants signing informed consent, according to Law no.12/2005, DL no.131/2014 and the Norm 015/2013 of the Directorate-General of Health (DGS), following the Tenets of the Helsinki Declaration. Samples were anonymized following the European Union General Data Protection Regulation (GDPR - EU 2016/679) and the Portuguese Law (Law no.58/2019).

Sociodemographic data, including age, educational level, marital status and profession were obtained by filling in the questionnaire that included the psychological assessment provided by the psychology team members.

This is the first study assessing changes in biomarkers and psychological symptoms in adults with cancer, in particular related to clown performances in treatment rooms. This is a pilot study, in which 64 women were analyzed: experimental group (EG; n=36; HCs intervention plus hosting conditions) versus control group (CG; n=28; hosting conditions). It is important to stress out the novelty of this work, in which a set of well-being biomarkers is implemented, in correlation with psychological evaluation including cognitive function, besides emotional states, all evaluated by cluster analysis.

The psychological assessment protocol covered affective, cognitive and satisfaction aspects of the intervention, in the form of both quantitative and qualitative data. The affective dimension was assessed in both groups using the Emotional States Perception Scale (PESS, with lower values corresponding to a better emotional state), the Positive Affectivity and Negative Affectivity Scale (PANAS, with higher and lower values, respectively, better affectivity), the Cognitive and Affective Mindfulness Scale-Revised (CAMS-R, a measure of attention, tolerance and acceptance of the present moment, with higher values corresponding to better results in these aspects). The cognitive dimension was assessed using the Clock-Drawing Test (CDT, with higher values corresponding to better cognitive functioning). The CDT, as a neuropsychological measure, assesses visuospatial, visuoconstructive and visuomotor abilities. It also involves other cognitive functions, including language/comprehension, memory, attention and executive functions (planning, organization, simultaneous processing, self-monitoring). It is also used as a brief cognitive screening test.

In the post-test, the EG was also assessed in terms of the importance and satisfaction attributed to the HCs intervention, as well as free-explanation testimonies, based on an open question, which finalized the assessment protocol in this group.

Concerning statistical analysis, primarily the qualitative data were described by its absolute and relative frequency while mean ± standard deviation and median [Quartile 1; Quartile3] were presented for quantitative data.

A factorial repeated measures ANOVA was applied in order to evaluate either the effect of evaluation moments and group interaction, and the main effect of the repeated measure (although some variables have presented normality deviations on their residuals, that fact did not have a significant impact on lowering power on those analysis). Moreover, bivariate comparisons between evaluations in each group were performed either using a Student's t-test for paired samples or a Wilcoxon test, according to sample distribution, and between groups for each time point using an independent samples t-test or a Mann-Whitney U-test using the same criteria. Pearson and Spearman rank order correlations between pre-test and post-test difference in biomarkers and psychological characteristics were also obtained for each group, and they were evaluated according to each data distribution. Furthermore, the differences of the changes in time of the variables were evaluated in function of the age and educational level of the patients between the two groups using a repeated measures ANOVA considering those as factors in a full factorial model.

These analyses were performed in IBM SPSS, version 25, and were analyzed at a 5% significance level (at a 10% significance level concerning Pearson and Spearman rank order correlations).

In order to assess association between biomarkers and psychological characteristics, cluster analyses using a Manhattan distance with single linkage were performed in Orange version 3.28.0 and the dendrograms obtained were presented.

ELIGIBILITY:
Inclusion Criteria:

* Adult women with cancer undergoing chemotherapy in the ambulatory hospital

Exclusion Criteria:

* Patients with head and neck cancer
* Having their first or last chemotherapy session
* Receiving chemotherapy orally or via lumbar puncture
* Presenting with any cognitive or language impairment that would prevent their understanding of the study and assessment or that could predictably interfere the levels of biomarkers evaluated

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only women were included in order to avoid gender based bias, concerning well being biomarkers.
  Participant eligibility is based on self-representation of gender identity.
Enrollment: 64 (Actual)
Dates: Start 2020-08-21 (Actual); Primary Completion 2020-08-28 (Actual); Study Completion 2020-08-28 (Actual)

PRIMARY OUTCOMES:
Oxytocin levels (saliva) | Basal and after ~ 90 minutes, during the chemotherapy treatment session
  Saliva collection for the biomarkers analysis was followed by psychological assessment, both at baseline (pre-test) and after ~90 minutes (post-test).
  The procedure was similar for all participants, considering the HCs intervention duration of 15 minutes performed between the baseline (pre-test) and after ~90 minutes (post-test) in the EG.
  Saliva collections were performed by the participants themselves, following instructions and using Saliva Collection Aid Salimetrics (5016.02-SAL), and stored at 4°C.
  The evaluation of oxytocin levels was performed by using the colorimetric competitive enzyme immunoassay ELISA kit ADI-900-153A (Enzo Life Sciences). Oxytocin extraction was required prior to ELISA, using SPE columns, acetonitrile and trifluoroacetic acid, according to manufacturers' instructions. All the samples were analyzed in duplicate, the saliva oxytocin content was expressed in pg/mL, determined by plotting the optical density of each sample against the standard curve.
Cortisol levels (saliva) | Basal and after ~ 90 minutes, during the chemotherapy treatment session
  Saliva collection for the biomarkers analysis was followed by psychological assessment, both at baseline (pre-test) and after ~90 minutes (post-test).
  The procedure was similar for all participants, considering the HCs intervention duration of 15 minutes performed between the baseline (pre-test) and after ~90 minutes (post-test) in the EG.
  Saliva collections were performed by the participants themselves, following instructions and using Saliva Collection Aid Salimetrics (5016.02-SAL). The samples were collected according to the schedule as described above and stored at 4°C.
  The evaluation of cortisol levels was performed by using the colorimetric competitive enzyme immunoassay ELISA kit ADI-900-071 (Enzo Life Sciences). The samples were thawed and centrifuged for immediate immunoassay processing in duplicate. A standard curve was used to estimate the cortisol content (pg/mL).
Serotonin levels (saliva) | Basal and after ~ 90 minutes, during the chemotherapy treatment session
  Saliva collection for the biomarkers analysis was followed by psychological assessment, both at baseline (pre-test) and after ~90 minutes (post-test).
  The procedure was similar for all participants, considering the HCs intervention duration of 15 minutes performed between the baseline (pre-test) and after ~90 minutes (post-test) in the EG.
  Saliva collections were performed by the participants themselves, following instructions and using Saliva Collection Aid Salimetrics (5016.02-SAL) and stored at 4°C.
  In the serotonin determination, samples were concentrated by lyophilization. The samples were frozen in liquid nitrogen and then processed in a freeze dryer. The serotonin ELISA assay was performed using a colorimetric competitive enzyme immunoassay (ADI-900-175 (Enzo Life Sciences)) kit, following to manufacturers' directions. The optical density (OD) was red at λ=405nm and the serotonin content (ng/mL) was determined by plotting OD of each sample against the standard curve.
ATP levels (saliva) | Basal and after ~ 90 minutes, during the chemotherapy treatment session
  Saliva collection for the biomarkers analysis was followed by psychological assessment, both at baseline (pre-test) and after ~90 minutes (post-test).
  The procedure was similar for all participants, considering the HCs intervention duration of 15 minutes made between the baseline (pre-test) and after ~90 minutes (post-test) in the EG.
  Saliva collections were performed by the participants themselves, following instructions and using Saliva Collection Aid Salimetrics (5016.02-SAL), according to the schedule described and stored at 4°C.
  The assessment of the saliva ATP levels was performed using a bioluminescent assay (ATP Bioluminescence Assay Kit HS II, Roche Diagnostics). This technique uses the ATP dependence on oxidation catalyzed by luciferase and allows the measurement of extremely low concentrations of ATP (up to 10-15 mol) in the saliva samples. The protein concentration was assayed by the Bradford method, and ATP levels were expressed normalized to that concentration.

SECONDARY OUTCOMES:
Positive Affect (PA) | Basal and after ~ 90 minutes, during the chemotherapy treatment session
  Psychological assessment was performed after saliva collection, both at baseline (pre-test) and after ~90 minutes (post-test).
  The procedure was similar for all participants, considering the HCs intervention duration of 15 minutes performed between the baseline (pre-test) and after ~90 minutes (post-test) in the EG.
  Affectivity was assessed by the Positive and Negative Affect Schedule (PANAS). The PANAS has two independent subscales with five items each. Responses are in a Likert scale and can vary from 1 ("Nothing or very slightly") to 5 ("Extremely"). The PANAS can measure affective and mood states in the moment. Higher values in positive affect (PA) and lower values in negative affect (NA) correspond, respectively, to a better affectivity. The Portuguese adaptation showed good psychometric properties, internal consistency (Cronbach's alpha =0.86 for PA) and 0.89 for NA) and structural validity through Confirmatory Factor Analysis.
Negative Affect (NA) | Basal and after ~ 90 minutes, during the chemotherapy treatment session
  Psychological assessment was performed after saliva collection, both at baseline (pre-test) and after ~90 minutes (post-test).
  The procedure was similar for all participants, considering the HCs intervention duration of 15 minutes performed between the baseline (pre-test) and after ~90 minutes (post-test) in the EG.
  Affectivity was assessed by the Positive and Negative Affect Schedule (PANAS). The PANAS has two independent subscales with five items each. Responses are in a Likert scale and can vary from 1 ("Nothing or very slightly") to 5 ("Extremely"). The PANAS can measure affective and mood states in the moment. Higher values in positive affect (PA) and lower values in negative affect (NA) correspond, respectively, to a better affectivity. The Portuguese adaptation showed good psychometric properties, internal consistency (Cronbach's alpha =0.86 for PA) and 0.89 for NA) and structural validity through Confirmatory Factor Analysis.
Emotional States (PESS) | Basal and after ~ 90 minutes, during the chemotherapy treatment session
  Psychological assessment was performed after saliva collection, both at baseline (pre-test) and after ~90 minutes (post-test).
  The procedure was similar for all participants, considering the HCs intervention duration of 15 minutes performed between the baseline (pre-test) and after ~90 minutes (post-test) in the EG.
  Emotional States were assessed by the Perception of Emotional States Scale (PESS), based on semantic differential scales and consisting of 8 pairs of opposite adjectives separated by 7 positions (e.g., calm/nervous; happy/sad). These pairs were selected because they represent emotional states, different from the affective states assessed by PANAS. Lower ratings correspond to a better emotional state.
Cognitive and Affective Mindfulness (CAMS-R) | Basal and after ~ 90 minutes, during the chemotherapy treatment session
  Psychological assessment was performed after saliva collection, both at baseline (pre-test) and after ~90 minutes (post-test).
  The procedure was similar for all participants, considering the HCs intervention duration of 15 minutes performed between the baseline (pre-test) and after ~90 minutes (post-test) in the EG.
  Cognitive and Affective Mindfulness was measured by the Cognitive and Affective Mindfulness Scale-Revised (CAMS-R), having 9 items rated to a 4-point Likert scale, ranging from 1 (Not at all) to 4 (A lot) and measures mindfulness qualities of attention, tolerance and acceptance of the present moment, with higher values corresponding to better results. For the present study, only 6 items were considered, because of the need to make the psychological assessment as brief as possible so that a minimum interference with ambulatory sessions functioning would occur and respecting the patient's availability could be ensured.
Cognitive functioning (CDT) | Basal and after ~ 90 minutes, during the chemotherapy treatment session
  Psychological assessment was performed after saliva collection, both at baseline (pre-test) and after ~90 minutes (post-test).
  The procedure was similar for all participants, considering the HCs intervention duration of 15 minutes performed between the baseline (pre-test) and after ~90 minutes (post-test) in the EG.
  Cognitive functioning was assessed by the Clock-Drawing Test (CDT, with higher values corresponding to better cognitive functioning). The CDT measures visuospatial, visuoconstructive and visuomotor capabilities. This test also evaluates other cognitive functions, including language/understanding, memory, attention and executive functions (planning, organization, simultaneous processing, self-monitoring). It is commonly used as a brief cognitive screening test. The Portuguese version of the 18-point quantitative scoring system was used.
Satisfaction with HCs' intervention | After ~ 90 minutes from basal, during the chemotherapy treatment session
  Satisfaction with HCs' intervention was evaluated in EG through two single items: (1) "Do you think this type of interventions in the hospital is important?", answered on a 4-point Likert scale (ranging between "Very important" and "Nothing important"); and (2) "How satisfied are you with the intervention of the HCs that you just saw?" answered in a 5-point Likert scale (ranging between "Very Satisfied" and "Very Unsatisfied").

CONTACTS AND LOCATIONS:
Overall Officials: Manuela Grazina, Principal Investigator — University of Coimbra
Locations (3):
- Portugal (3):
  - Instituto Português de Oncologia de Coimbra Francisco Gentil, E.P.E., Coimbra
  - University of Coimbra - Faculty of Psichology, Coimbra
  - University of Coimbra - Laboratory of Mitochondrial Biomedicine and Theranostics, Coimbra

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tuckman, B.W., 2012. Manual de investigação em educação: Metodologia para conceber e realizar o processo de investigação científica, 2nd ed. Fundação Calouste Gulbenkian.
- [Background] Galinha, I.C., Pereira, C.R., Esteves, F., 2014. Versão reduzida da escala portuguesa de afeto positivo e negativo - PANAS-VRP: Análise fatorial confirmatória e invariância temporal [Short-Form of the Portuguese version of the positive and negative affect schedule - PANAS-Port-VRP: Confirmatory factorial analysis and temporal invariance]. Psicologia. 28 (1), 53-65. http://scielo.pt/scielo.php?script=sci_arttext&pid=S0874-20492014000100005&lng=pt&tlng=pt.
- [Background] Teixeira, R.J., Ferreira, G., Pereira, M.G., 2017. Portuguese validation of the Cognitive and Affective. Mindfulness & Compassion. 2, 3-8. https://doi.org/10.1016/J.MINCOM.2017.03.001.
- [Background] Santana I, Duro D, Freitas S, Alves L, Simoes MR. The Clock Drawing Test: Portuguese norms, by age and education, for three different scoring systems. Arch Clin Neuropsychol. 2013 Jun;28(4):375-87. doi: 10.1093/arclin/act016. Epub 2013 Mar 21. PMID 23518874
- [Background] Casellas-Grau A, Ochoa C, Lleras De Frutos M, Flix-Valle A, Rosales A, Gil F. Perceived changes in psychological and physical symptoms after hospital clown performances in a cancer setting. Arts Health. 2021 Jun;13(2):189-203. doi: 10.1080/17533015.2020.1744172. Epub 2020 Mar 29. PMID 32223531
- [Background] Ferreira AC, Osorio FL. Peripheral oxytocin concentrations in psychiatric disorders - A systematic review and methanalysis: Further evidence. Prog Neuropsychopharmacol Biol Psychiatry. 2022 Jul 13;117:110561. doi: 10.1016/j.pnpbp.2022.110561. Epub 2022 Apr 21. PMID 35461971
- [Background] Chojnowska S, Ptaszynska-Sarosiek I, Kepka A, Knas M, Waszkiewicz N. Salivary Biomarkers of Stress, Anxiety and Depression. J Clin Med. 2021 Feb 1;10(3):517. doi: 10.3390/jcm10030517. PMID 33535653
- [Background] Matsunaga M, Ishii K, Ohtsubo Y, Noguchi Y, Ochi M, Yamasue H. Association between salivary serotonin and the social sharing of happiness. PLoS One. 2017 Jul 6;12(7):e0180391. doi: 10.1371/journal.pone.0180391. eCollection 2017. PMID 28683075
- [Background] Picard M, McEwen BS, Epel ES, Sandi C. An energetic view of stress: Focus on mitochondria. Front Neuroendocrinol. 2018 Apr;49:72-85. doi: 10.1016/j.yfrne.2018.01.001. Epub 2018 Jan 12. PMID 29339091
- [Background] Steckl AJ, Ray P. Stress Biomarkers in Biological Fluids and Their Point-of-Use Detection. ACS Sens. 2018 Oct 26;3(10):2025-2044. doi: 10.1021/acssensors.8b00726. Epub 2018 Oct 16. PMID 30264989
- [Background] Feldman R. The Neurobiology of Human Attachments. Trends Cogn Sci. 2017 Feb;21(2):80-99. doi: 10.1016/j.tics.2016.11.007. Epub 2016 Dec 30. PMID 28041836
- [Background] Tijssen, P. (1985). Practice & Theory of Enzyme Immunoassays. Elsevier, Amsterdam.
- [Background] Kruger NJ. The Bradford method for protein quantitation. Methods Mol Biol. 1994;32:9-15. doi: 10.1385/0-89603-268-X:9. No abstract available. PMID 7951753
- [Background] Bioluminescence and chemiluminescence. Methods Enzymol. 1978;57:1-653. No abstract available. PMID 732586
- [Background] Babins L, Slater ME, Whitehead V, Chertkow H. Can an 18-point clock-drawing scoring system predict dementia in elderly individuals with mild cognitive impairment? J Clin Exp Neuropsychol. 2008 Feb;30(2):173-86. doi: 10.1080/13803390701336411. PMID 18938669